CLINICAL TRIAL: NCT03887715
Title: A Prospective, Multi-center, Randomized Controlled Blinded Trial Demonstrating the Safety and Effectiveness of VNS Therapy® System as Adjunctive Therapy Versus a No Stimulation Control in Subjects With Treatment-Resistant Depression
Acronym: RECOVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LND-300
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression
Keywords: VNS; Depression; TRD
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of active stimulation vs. no stimulation for 12 months post randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Central Rater and sponsor are blinded in the RCT phase. Sites will need to have an unblinded programmer who is only programming the device and not collecting outcomes data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active (Active Comparator): Group will have VNS activated 2 weeks post implant.
  Interventions: Device: Vagus Nerve Stimulation (VNS)
- Control (Sham Comparator): Group will be implanted with VNS but device is not activated for the first 12 months. After 12 months, this group can receive stimulation.
  Interventions: Device: Vagus Nerve Stimulation (VNS)

INTERVENTIONS:
Device: Vagus Nerve Stimulation (VNS) — VNS is an implantable device that delivers stimulation to the vagal nerve.
  Other Names: VNS

SUMMARY:
Objectives of this study are to determine whether active VNS Therapy treatment is superior to a no stimulation control in producing a reduction in baseline depressive symptom severity, based on multiple depression scale assessment tools at 12 months from randomization.

DETAILED DESCRIPTION:
A prospective, multi-center, randomized, controlled, blinded trial of subjects implanted with VNS Therapy. Active treatment and no stimulation control are randomized, at least two weeks after implantation and observed for 12-months.

After completing the 12 month endpoint in the RCT portion of the study, all RECOVER subjects will transition into the prospective, open-label, longitudinal portion of the study. Subjects in the control arm of RECOVER will be activated after completing the 12 month endpoint.

After completion of enrollment in the RCT portion or meeting of interim success criterion (whichever comes first), up to 5,800 new subjects may enroll directly into the open-label,prospective, longitudinal study. These subjects will participate in the study for approximately 5 years.

The study has been designed in accordance with The Centers for Medicare and Medicaid Services coverage with evidence development (CED) decision entitled "Decision Memo for Vagus Nerve Stimulation (VNS) for Treatment Resistant Depression (TRD) (CAG-00313R2).

ELIGIBILITY:
Inclusion Criteria:

The patient must be in a major depressive disorder (MDD) episode for ≥ two years or have had at least four episodes of MDD, including the current episode.

The patient's depressive illness meets a minimum criterion of four prior failed treatments of adequate dose and duration as measured by a tool designed for this purpose.

The patient is experiencing a major depressive episode (MDE) as measured by a guideline recommended depression scale assessment tool on two visits, within a 45-day span prior to implantation of the VNS device.

Patients must maintain a stable medication regimen for at least four weeks before device implantation.

Exclusion Criteria:

Current or lifetime history of psychotic features in any MDE;

Current or lifetime history of schizophrenia or schizoaffective disorder;

Current or lifetime history of any other psychotic disorder;

Current or lifetime history of rapid cycling bipolar disorder;

Current secondary diagnosis of delirium, dementia, amnesia, or other cognitive disorder;

Current suicidal intent; or

Treatment with another investigational device or investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6800 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale (MADRS) Rate of Response | 12 months post randomization
  The rate of response defined as person months of response/total months of study participation where response is at least a 50% reduction from baseline in MADRS total score. Subjects discontinuing the study before the endpoint assessment will be considered as non-responders for each successive month after discontinuance.
Montgomery Åsberg Depression Rating Scale (MADRS) Time to First response | Baseline up to 12 Months
  Time from randomization to the first observed MADRS response.
Montgomery Åsberg Depression Rating Scale (MADRS) Time to First Remission | Baseline up to 12 Months
  Time from randomization to the first observed MADRS remission.
Montgomery Åsberg Depression Rating Scale (MADRS) Duration of Response | Baseline up to 12 Months
  Duration of MADRS response, defined as the number of consecutive months from first observed MADRS response to the first assessment of MADRS response relapse.
Montgomery Åsberg Depression Rating Scale (MADRS) Rate of Remission | Baseline up to 12 Months
  The rate of remission is defined as total number of months in remission divided by total months of expected study participation. Subjects discontinuing the study before the endpoint assessment will be considered as non-in-remission for each successive month after discontinuance
Montgomery Åsberg Depression Rating Scale (MADRS) Maximum duration of Response | Baseline up to 12 Months
  Maximum duration of MADRS response, defined as the maximum number of consecutive months in response (only for subjects experiencing MADRS response).
Montgomery Åsberg Depression Rating Scale (MADRS) Duration of Remission | Baseline up to 12 Months
  Duration of MADRS remission, defined as the number of consecutive months from first observed MADRS remission to the first assessment of MADRS remission relapse (defined score > 20).
Montgomery Åsberg Depression Rating Scale (MADRS) Maximum duration of Remission | Baseline up to 12 Months
  Maximum duration of MADRS remission, defined as the maximum number of consecutive months in remission (only for subjects experiencing MADRS remission).
Assess all Adverse Events | Implant to 12 Months
  All adverse events, with a focus on device or procedure-related serious adverse events.
WHO Disability Assessment Schedule (WHODAS) Changes in scores over time | Baseline to 12 Months
Health Outcome Scale (EQ-5D-L) Changes in scores over time | Baseline to 12 Months
Clinical Global Impressions Scale - Improvement (CGI-I) Response | 12 months post randomization
  A CGI-I score ≤ 2 at 12 months from randomization. Subjects discontinuing the study before the 12 months assessment will be considered as not in response for each successive month after discontinuance.
Sheehan Suicidality Tracking Scale (S-STS) Changes in Suicidality | Implant to 12 Months
  Suicide attempts as measured by items #10 & #12 in S-STS scale

CONTACTS AND LOCATIONS:
Overall Officials: Charles Conway, MD, Principal Investigator — Washington University School of Medicine
Locations (98):
- United States (98):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UAB Huntsville Regional Medical Center, Huntsville, Alabama
  - Access Multi Specialty Medical Clinic, Inc, Burlingame, California
  - CMB Clinical Trials, Colton, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Kaizen Brain Center, La Jolla, California
  - Keck Hospital of USC, Los Angeles, California
  - University of California San Diego, San Diego, California
  - SF-CARE, Inc., San Rafael, California
  - Syrentis Clinical Research, Santa Ana, California
  - Sunrise Research Institute, Boca Raton, Florida
  - Mindful Behavioral Health, Boca Raton, Florida
  - Medycal Research, Inc, Brooksville, Florida
  - Galiz Research LLC, Hialeah, Florida
  - Florida Behavioral Psych, Largo, Florida
  - Segal Trials Corporate, Lauderhill, Florida
  - Central Miami Medical Institute, LLC, Miami, Florida
  - Clintex Research Group, Inc., Miami, Florida
  - Research Center Of Florida, Inc, Miami, Florida
  - Ocean Blue Medical Research Center, Miami Springs, Florida
  - APG Research, LLC, Orlando, Florida
  - Nova Psychiatry Inc., Orlando, Florida
  - Florida Center for TMS, Orlando, Florida
  - Millenia Psychiatry & Research, Inc, Orlando, Florida
  - Quantum Laboratories Inc., Pompano Beach, Florida
  - Advanced Mental Health Care Inc., Royal Palm Beach, Florida
  - Florida Center for TMS, Saint Augustine, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Psychiatric Specialty Center, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta University, Augusta, Georgia
  - PACT Atlanta LLC, Decatur, Georgia
  - IACT Health, Grayson, Georgia
  - Psych Atlanta, Marietta, Georgia
  - Pearl Health Clinic, Ammon, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Joliet Center For Clinical Research, Joliet, Illinois
  - AMR- Baber Research, Inc., Naperville, Illinois
  - Psychiatric Medicine Associates, LLC, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Neuroscience Research Institute, Winfield, Illinois
  - Advanced Research Institute, Inc., Indianapolis, Indiana
  - Beacon Medical Group Behavioral Health, South Bend, Indiana
  - University Of Kansas Cancer Center, Kansas City, Kansas
  - Sheppard Pratt Health System, Inc., Baltimore, Maryland
  - Clinical Insights, Glen Burnie, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Precise Research Centers, Flowood, Mississippi
  - Andrew Bishop, MD, Jackson, Mississippi
  - University of Missouri, Columbia, Missouri
  - Psychiatric Care and Research, O'Fallon, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Healthy Perspective, Nashua, New Hampshire
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - University of New Mexico - Psychiatric Center, Albuquerque, New Mexico
  - Dent Neurological Institute, Amherst, New York
  - Erie County Medical Center/State University of New York (SUNY) at Buffalo Affiliate, Buffalo, New York
  - Trinity Medical, Lewiston, New York
  - Hapworth Research Inc., New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - State University Of New York Upstate Medical University, Syracuse, New York
  - ManuMind Interventional Psychiatry, Woodbury, New York
  - The Center for Neuropsychiatry and Brain Stimulation (CNBS) ARC Health, Cary, North Carolina
  - Mindpath Care Centers, Raleigh, North Carolina
  - Wake Forest University Health Science, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Signature Research Associates, Inc., Fairlawn, Ohio
  - Charak Center for Health and Wellness, Garfield Heights, Ohio
  - NPC Research, Oklahoma City, Oklahoma
  - Rivus Wellness & Research Institute, Oklahoma City, Oklahoma
  - University of Oklahoma School of Community Medicine, Tulsa, Oklahoma
  - Scranton Medical Institutes, Moosic, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Neuroscience and TMS Treatment Center, Brentwood, Tennessee
  - UT Health Austin, Mulva Clinic for the Neurosciences, Austin, Texas
  - BioBehavioral Research of Austin, Austin, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Texas Tech University Health Science Center, El Paso, Texas
  - The University Of Texas Medical School At Houston - UT Center Of Excellence On Mood Disorders, Houston, Texas
  - Houston Clinical Trials, Houston, Texas
  - Northpointe Psychiatry, Lewisville, Texas
  - Rise Clinical Research, LLC, Missouri City, Texas
  - The University of Utah, Salt Lake City, Utah
  - Neuropsychiatric Associates, Plc, Woodstock, Vermont
  - Carilion Clinic, Roanoke, Virginia
  - Center For Anxiety and Depression, Mercer Island, Washington
  - Seattle Neuropsychiatric Treatment Center, Seattle, Washington
  - Marshall University Joan C. Edwards School of Medicine, Huntington, West Virginia
  - West Virginia Clinical and Translational Science Institute, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aaronson ST, Conway CR, Gordon C, Lee YL, George MS, Zajecka J, Riva-Posse P, Dunner DL, Macaluso M, Rosenquist PB, Mickey BJ, Sheline YI, Hristidis VC, Brown H, Kriedt CL, Tran Q, Bunker MT, Sackeim HA, Rush AJ. Prognostic and Prescriptive Predictors of Treatment Response to Adjunctive VNS Therapy in Major Depressive Disorder: A RECOVER Trial Report. J Clin Psychiatry. 2025 Jul 14;86(3):25m15850. doi: 10.4088/JCP.25m15850. PMID 40673907
- [Derived] de Leon VC, Allen RM, Quevedo J, Riva-Posse P, Aaronson ST, Berger MA, Zajecka J, Banov MD, Manu LM, Sheline YI, Farrington J, Eloge JC, Beard J, Kriedt CL, Gott BM, Brown H, Bunker MT, Lee YL, Rush AJ, Sackeim HA, Conway CR. Suicide characteristics in patients with marked treatment-resistant major depressive disorder: A RECOVER trial report. J Affect Disord. 2025 Apr 1;374:619-629. doi: 10.1016/j.jad.2024.12.072. Epub 2024 Dec 24. PMID 39722333
- [Derived] Conway CR, Aaronson ST, Sackeim HA, Duffy W, Stedman M, Quevedo J, Allen RM, Riva-Posse P, Berger MA, Alva G, Malik MA, Dunner DL, Cichowicz I, Luing H, Zajecka J, Nahas Z, Mickey BJ, Kablinger AS, Kriedt CL, Bunker MT, Lee YL, Shy O, Majewski S, Olin B, Tran Q, Rush AJ. Clinical characteristics and treatment exposure of patients with marked treatment-resistant unipolar major depressive disorder: A RECOVER trial report. Brain Stimul. 2024 Mar-Apr;17(2):448-459. doi: 10.1016/j.brs.2024.03.016. Epub 2024 Apr 2. PMID 38574853
- See also: CMS Decision Memo for Vagus Nerve Stimulation (VNS) for Treatment Resistant Depression — https://www.cms.gov/medicare-coverage-database/details/nca-decision-memo.aspx?NCAId=292